CLINICAL TRIAL: NCT05712837
Title: Efficacy of 25% Trichloroacetic Acid Peel Versus 30% Salicylic Acid Peel in Mild to Moderate Acne Vulgaris
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Combined Military Hospital Abbottabad (Other)
Responsible Party: Principal Investigator, Dr kiran gul, principal investigator, Combined Military Hospital Abbottabad
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMHAtd-ETH-15-Derm-22
Record Dates: First submitted 2023-01-18; First posted 2023-02-06 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-01

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Trichloroacetic Acid; Salicylic Acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A 25% TCA (Active Comparator): 25% TCA peel Patients of group A were treated with 25% TCA peel and patients at 2-week intervals for a total of 12 weeks. Clinical evaluation was done at the end of therapy after 12-weeks of treatment.
  Interventions: Drug: 25% TRICHLOROACETIC ACID
- Group B 30% SALICYLIC ACID (Active Comparator): 30% SA peels Patients of group B were treated with 30 % salicylic acid peel and patients at 2 weeks interval for a total of 12 weeks.clinical evaluation was done at the end of therapy after 12 weeks of treatment
  Interventions: Drug: 30% salicylic acid

INTERVENTIONS:
Drug: 25% TRICHLOROACETIC ACID — Patients of group A were treated with 25% TCA peel and patients at 2-week intervals for a total of 12 weeks. Clinical evaluation was done at the end of therapy after 12-weeks of treatment.
  Other Names: Peeling agent
  Arms: Group A 25% TCA
Drug: 30% salicylic acid — Patients of group B were treated with 30 % salicylic acid peel and patients at 2 weeks interval for a total of 12 weeks.clinical evaluation was done at the end of therapy after 12 weeks of treatment
  Other Names: Peeling agent
  Arms: Group B 30% SALICYLIC ACID

SUMMARY:
To compare the efficacy of 25% trichloroacetic acid peel versus 30% salicylic acid peel in mild to moderate acne vulgaris.

Study Design: Randomized Control Trial. Place And Duration of Study: Department of Dermatology, CMH Abbottabad from 01 Jun 2022 to 30th Nov, 2022.

Methodology: A total of 60 patients presented with mild or moderate acne vulgaris were randomized into two groups comprising 30 patients in each group and treated with either the TCA peel or the SA peel at 2-week intervals for 12 weeks. Patients in Group A were treated with 25% TCA peel whereas patients in Group B were treated with 30% SA peel. At the end of therapy after 12 weeks, evaluation of active acne was done by individual lesion counts (comedones, papules and pustules) and calculation of the Michaelsson acne score (MAS).

ELIGIBILITY:
Inclusion Criteria:

* Patients with mild or moderate facial acne vulgaris presented in dermatology opd

Exclusion Criteria:

* Patients with grade III or IV acne vulgaris
* patients taking any acne medications or had taken oral or topical medications in the past 4 weeks
* pregnant female patients or nursing a baby
* patients with known hypersensitivity to the formulations used in the study or a history of photosensitivity
* hypertrophic scars, keloidal tendency, active or recurrent herpes simplex infection
* active dermatosis
* unrealistic expectations

Ages: 13 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Effectiveness of 25 % trichloroacetic acid peel versus 30 % salicylic acid peel in the treatment of mild to moderate acne vulgaris | 12 weeks
  Michaelson acne scores (MAS) Michaelson acne scores (MAS) was used to measure the effectiveness of both peels

CONTACTS AND LOCATIONS:
Locations (1):
- Cmh abbottabad, Abbottābād, Kpk, Pakistan